CLINICAL TRIAL: NCT04035031
Title: Effects of SGLT-2 Inhibitor Dapagliflozin on Hormonal Glucose Regulation and Ketogenesis in Patients With Type 1 Diabetes - a Randomised, Placebo-controlled, Open-label, Cross-over Intervention Study
Brief Title: Effects of Dapagliflozin on Hormonal Glucose Homeostasis in Type 1 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CUI_002_01
Record Dates: First submitted 2019-07-24; First posted 2019-07-29 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Randomised, placebo-controlled, open-label, cross over intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Forxiga first, placebo second (Experimental): Forxiga followed by placebo
  Interventions: Drug: Forxiga 10mg; Drug: Placebo
- Placebo first, Forxiga second (Experimental): Placebo followed by forxiga
  Interventions: Drug: Forxiga 10mg; Drug: Placebo

INTERVENTIONS:
Drug: Forxiga 10mg — Forxiga™ 10mg, dapagliflozin 10mg, oral, once daily for 7 days (70 mg total)
  Other Names: Dapagliflozin
Drug: Placebo — Placebo tablets, starch, oral, once daily for 7 days (7 tablets total)

SUMMARY:
Inhibitors of sodium-dependent glucose-transporter 2 (including dapagliflozin) represent intensively investigated drugs in the field of diabetes. SGLT-2 inhibition limits glucose reabsorption in renal tubular cells, hereby increasing the amount of glucose excreted via urine in the hyperglycemic state. Its mechanisms of action are independent of insulin, the indispensable standard of care in Type 1 Diabetes (T1D). Several international diabetes experts highlighted the need for adjunct therapies in T1D.

Subcutaneous application of insulin is non-physiological. Most significant, subcutaneous insulin substitution does not address the bi-hormonal character of T1D. The loss of pancreatic beta cells and subsequent endogenous insulin production uncouples alpha cell derived glucagon secretion from its paracrine suppressor. Consequently, excess glucagon concentrations occur in the fasting and the postprandial state, which promotes hyperglycemia, requires higher doses of subcutaneous insulin, and promotes glycaemic variability.

Recent studies on SGLT-2 inhibition in T1D showed better glycemic control compared to placebo, whereas a higher risk for the development of diabetic ketoacidosis was observed. Knowledge about the underlying mechanisms is scarce. Studies showed that SGLT-inhibition increased Glucagon-like-peptide 1 (GLP-1) in T1D, an incretin hormone capable of suppressing glucagon. On the other side, total concentrations of ketone bodies were higher following SGLT-2 inhibition, irrespective of ongoing subcutaneous or intravenous insulin substitution. The present study aims to investigate the effect of SGLT-2 inhibitor dapagliflozin on hormonal regulators of glucose homeostasis and ketogenesis in T1D. The primary endpoint is the difference of GLP-1 during oral glucose tolerance test clamps (OGGTc). Secondary endpoints comprise total ketone body concentrations, free fatty acids, glucagon, and somatostatin during OGTTc and hyperinsulinemic, euglycemic clamps (HEC) following dapagliflozin and placebo. The study recruits male and female patients with T1DM in a randomized, open label, cross-over intervention study.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Duration of T1DM > 5 years
* Male or female sex
* Body mass index (BMI) between 20 and 29 kg/m2
* Adherence to safe contraception during the study and for 2 weeks after completion of the study protocol. Safe contraception comprises double barrier methods (hormonal contraception [like: oral contraceptive pills or intrauterine contraceptive devices] together with a mechanical barrier [like: condom, diaphragm]).

Exclusion Criteria:

* Contraindications to SGLT-2 inhibitors
* Contraindications to lactose
* Diagnosis of renal and/or hepatic dysfunction
* History of malignancy of any kind
* Intake of drugs influencing glucose homeostasis during the last three months (steroids, metformin, sulfonylureas, thiazolidinedione)
* Known or suspected non-compliance, drug or alcohol abuse.
* Inadequate vein status on both forearms
* Active smoker (defined as ≥1 or more cigarettes or nicotine-containing equivalents per day)
* Known pregnancy, positive plasma beta-HCG test prior to study inclusion or intention to become pregnant during the study period.
* Women who are breast feeding
* Lack of safe contraception
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2020-11-12 (Actual)

PRIMARY OUTCOMES:
Area under the curve for glucagon-like peptide I in oral glucose tolerance test clamp | From time-point 0 to 120 minutes during oral glucose tolerance test clamp, measurement every 15 minutes
  Glucagon-like peptide I will be measured in oral glucose tolerance test clamp following dapagliflozin and will be compared with concentrations measured following placebo. Active and inactivated glucagon like peptide I will be measured.
Area under the curve for glucagon-like peptide I in oral glucose tolerance test clamp | During visit 3 (day 7): From time-point 0 to 120 minutes during oral glucose tolerance test clamp, measurement every 15 minutes
  Glucagon-like peptide I will be measured in oral glucose tolerance test clamp following dapagliflozin and will be compared with concentrations measured following placebo. Active and inactivated glucagon like peptide I will be measured.
Area under the curve for glucagon-like peptide I in oral glucose tolerance test clamp | During visit 5 (day 31): From time-point 0 to 120 minutes during oral glucose tolerance test clamp, measurement every 15 minutes
  Glucagon-like peptide I will be measured in oral glucose tolerance test clamp following dapagliflozin and will be compared with concentrations measured following placebo. Active and inactivated glucagon like peptide I will be measured.

SECONDARY OUTCOMES:
Area under the curve for glucagon-like peptide I in euglycemic, hyperinsulinemic clamp | From time-point 0 to 120 minutes during euglycemic, hyperinsulinemic clamp, measurement every 15 minutes
  Glucagon-like peptide I will be measured in euglycemic, hyperinsulinemic clamp following dapagliflozin and will be compared with concentrations measured following placebo. Active and inactivated glucagon like peptide I will be measured.
Area under the curve for ketone body concentrations in euglycemic, hyperinsulinemic clamp following dapagliflozin compared with placebo | From time-point 0 to 120 minutes during euglycemic, hyperinsulinemic clamp, measurement every 15 minutes
  Ketone bodies will be measured in euglycemic, hyperinsulinemic clamp following dapagliflozin and will be compared with concentrations measured following placebo. Active and inactivated glucagon like peptide I will be measured.
Area under the curve for ketone body concentrations in oral glucose tolerance test clamp following dapagliflozin compared with placebo | From time-point 0 to 120 minutes during oral glucose tolerance test clamp, measurement every 15 minutes
  Ketone bodies will be measured in oral glucose tolerance test clamp following dapagliflozin and will be compared with concentrations measured following placebo. Active and inactivated glucagon like peptide I will be measured.
Area under the curve for free fatty acids in euglycemic, hyperinsulinemic clamp following dapagliflozin compared with placebo | From time-point 0 to 120 minutes during euglycemic, hyperinsulinemic clamp, measurement every 15 minutes
  Free fatty acids will be measured in euglycemic, hyperinsulinemic clamp following dapagliflozin and will be compared with concentrations measured following placebo. Active and inactivated glucagon like peptide I will be measured.
Area under the curve for free fatty acids in oral glucose tolerance test clamp following dapagliflozin compared with placebo | From time-point 0 to 120 minutes during oral glucose tolerance test clamp, measurement every 15 minutes
  Free fatty acids will be measured in oral glucose tolerance test clamp following dapagliflozin and will be compared with concentrations measured following placebo. Active and inactivated glucagon like peptide I will be measured.
Area under the curve for glucagon in euglycemic, hyperinsulinemic clamp following dapagliflozin compared with placebo | From time-point 0 to 120 minutes during euglycemic, hyperinsulinemic clamp, measurement every 15 minutes
  Glucagon will be measured in euglycemic, hyperinsulinemic clamp following dapagliflozin and will be compared with concentrations measured following placebo. Active and inactivated glucagon like peptide I will be measured.
Area under the curve for glucagon in oral glucose tolerance test clamp following dapagliflozin compared with placebo | From time-point 0 to 120 minutes during oral glucose tolerance test clamp, measurement every 15 minutes
  Glucagon will be measured in oral glucose tolerance test clamp following dapagliflozin and will be compared with concentrations measured following placebo. Active and inactivated glucagon like peptide I will be measured.
Area under the curve for somatostatin in euglycemic, hyperinsulinemic clamp following dapagliflozin compared with placebo | From time-point 0 to 120 minutes during euglycemic, hyperinsulinemic clamp, measurement every 15 minutes
  Somatostatin will be measured in euglycemic, hyperinsulinemic clamp following dapagliflozin and will be compared with concentrations measured following placebo. Active and inactivated glucagon like peptide I will be measured.
Area under the curve for somatostatin in oral glucose tolerance test clamp following dapagliflozin compared with placebo | From time-point 0 to 120 minutes during oral glucose tolerance test clamp, measurement every 15 minutes
  Somatostatin will be measured in oral glucose tolerance test clamp following dapagliflozin and will be compared with concentrations measured following placebo. Active and inactivated glucagon like peptide I will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Laimer, Prof. MD, Principal Investigator — Department of Diabetes, Endocrinology, Clinical Nutrition and Metabolism, University Clinics Bern, Inselspital, Bern, Switzerland
Locations (1):
- Department of Diabetes, Endocrinology, Nutritional Medicine and Metabolism, Inselspital, Bern University Hospital, University of Bern, Bern, Switzerland, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
According to Swiss National Fund (SNF) policy on Open Research Data, Data will be uploaded to an open data registry.
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Derived] Gubeli A, Steiner N, Limacher A, Mathis D, Melmer A, Laimer M. Dapagliflozin's impact on hormonal regulation and ketogenesis in type 1 diabetes: a randomised controlled crossover trial. Diabetologia. 2025 Oct;68(10):2116-2125. doi: 10.1007/s00125-025-06481-9. Epub 2025 Jul 9. PMID 40629004